CLINICAL TRIAL: NCT04988321
Title: Theta Burst Brain Stimulation in Diabetic Neuropathy Patients With Neuropathic Pain: Investigating Neural Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20021531
Record Dates: First submitted 2021-07-23; First posted 2021-08-03 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: transcranial magnetic stimulation; non-invasive brain stimulation
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary motor cortex (M1) (Active Comparator): Stimulation of the M1
  Interventions: Procedure: Prolonged continuous theta burst stimulation (pcTBS)
- Dorsolateral prefrontal cortex (DLPFC) (Active Comparator): Stimulation of the DLPFC
  Interventions: Procedure: Prolonged continuous theta burst stimulation (pcTBS)

INTERVENTIONS:
Procedure: Prolonged continuous theta burst stimulation (pcTBS) — Non-invasive brain stimulation (transcranial magnetic stimulation or TMS) which consists of a stimulating coil being held over the head. When this coil delivers a painless magnetic pulse, it feels like a quick, light tap on the head. Two different coils will be used to perform TMS. One coil will be used to determine stimulation parameters for the pcTBS protocol. The second coil will be used to implement pcTBS, which is a repetitive non-invasive brain stimulation protocol which feels like many quick, light taps on the head. Participants will receive two procedures during one session, one with active stimulation and one with inactive stimulation.

SUMMARY:
The purpose of the study is to determine the effects of a newer form of non-invasive brain stimulation (called transcranial magnetic stimulation or TMS) as a treatment in patients with painful diabetic neuropathy to examine its effects on their understanding of their pain experience.

DETAILED DESCRIPTION:
The proposed brain stimulation technique in this study is an investigational procedure that has not been approved by the U.S. FDA for treating pain linked to diabetic neuropathy, but it has been approved to treat depression. The study will use surveys to monitor how participant's body changes as their understanding of their pain experience changes. Participants will be randomized (like the flip of a coin) to receive brain stimulation at one of two brain regions which are involved in the processing and understanding of the pain experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type II Diabetes Mellitus.
* Age 18-75 years.
* Diagnosed by a Physician with diabetic neuropathy/ distal symmetric polyneuropathy/ diabetic polyneuropathy.
* Patients under physician care at Virginia Commonwealth University Health Systems in the Neurology Clinic/ Neurology Department and the Endocrinology Clinic
* Neuropathic pain for at least 3 months.
* Neuropathic pain signs and symptoms identified using Pain DETECT questionnaire.
* Current pain score ≥3 or higher (0='no pain' and 10='worst possible pain').
* Pain Medication dosage stable for at least 4 weeks

Exclusion Criteria:

* Non-neuropathic chronic pain
* Another concurrent cause of neuropathic pain
* Any history of epilepsy, drug-resistant migraine, and/or any presence of ferromagnetic implant, cardiac pacemakers, implanted insulin pumps, neurostimulators, cochlear implants and surgical clips or medical pumps.
* Limited English proficiency
* Pregnant patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Change in Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) score | Baseline to the end of the procedure, about 2.25 hours
  The QOL-DN is questionnaire is an instrument to assess quality of life in patients with diabetic polyneuropathy. It is comprised of 35 items and yields a Total QOL score.
Change in bodily and emotional perception of pain (BEEP) score | Baseline to the end of the procedure, about 2.25 hours
  The BEEP questionnaire is a self-report questionnaire measuring the impact of chronic pain on daily life. It has 23 items on a 0-5 Likert scale that assesses three pain dimensions, namely the emotional reaction to pain, the limitations to daily life caused by pain and the interference caused by pain in personal and social functioning. Responses are summed to yield a single BEEP score.

SECONDARY OUTCOMES:
Change in pain threshold - conditioned pain modulation (CPM) | Baseline to the end of the procedure, about 2.25 hours
  To measure CPM, brief amounts of slight pressure using a handheld pressure device will be applied to a location either on the forearm or leg where the patient reports a current absence of pain. An average index percent ratio will be calculated from the pressure device in kilopascals at which participants report the pressure was first perceived as painful during a baseline assessment and during an assessment when the participant's contralateral hand was placed in cold water. Change will be measured by subtracting CPM scores before and after the active procedure.
Change in pain threshold - Temporal Summation of Pain (TSP) | Baseline to the end of the procedure, about 2.25 hours
  To measure TSP, the same pressure using a handheld pressure device that was perceived as first painful will be applied to a location either on the forearm or leg where the patient reports a current absence of pain. This pressure will be applied repeatedly applied 10 times and participants will be asked to report their pain on a 0-10 scale where 0 is no pain and 10 is worst pain imaginable. Change will be measured by subtracting TSP scores before and after the active procedure.
Change in pain threshold - Offset Analgesia (OA) | Baseline to the end of the procedure, about 2.25 hours
  A Velcro strap tied to participants forearm connected to a device that transmits heat will be used to measure OA. Three different temperatures of mild heat will be applied. Participants will use a visual analog scale (VAS, no heat 0- extreme heat 10) to rate the intensity of the heat stimulus at each temperature. Minimal VAS ratings at the highest temperature will be subtracted from maximal VAS ratings at the lowest temperature to yield OA value. Change will be measured by subtracting OA values before and after the active procedure.
Change in cortical inhibition (CI) | Baseline to the end of the procedure, about 2.25 hours
  The amplitude the motor evoked potentials (MEPS) from two simultaneous pulses will be used to determine level of cortical inhibition.
Change in corticospinal excitability (CE) | Baseline to the end of the procedure, about 2.25 hours
  The amplitude the motor evoked potentials (MEPS) from a single pulse will be used to determine level of corticomotor excitability

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thakkar B, Peterson CL, Acevedo EO. Single Session Effects of Prolonged Continuous Theta Burst Stimulation Targeting Two Brain Regions on Pain Perception in Patients with Painful Diabetic Neuropathy: A Preliminary Study. J Integr Neurosci. 2024 Mar 7;23(3):54. doi: 10.31083/j.jin2303054. PMID 38538225